CLINICAL TRIAL: NCT01034358
Title: Comparison of Immune Response to the Human Papillomavirus Vaccine in Young Women With and Without Inflammatory Bowel Disease
Brief Title: Immune Response to the Human Papillomavirus Vaccine in Young Women With Inflammatory Bowel Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Jeanne Tung, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09-000485
Record Dates: First submitted 2009-12-10; First posted 2009-12-17 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-09

CONDITIONS: Inflammatory Bowel Disease; Uterine Cervical Dysplasia
Keywords: inflammatory bowel disease; Crohn disease; ulcerative colitis; Papillomavirus vaccines
MeSH Terms: conditions — Inflammatory Bowel Diseases; Uterine Cervical Dysplasia; Crohn Disease; Colitis, Ulcerative | interventions — Papillomavirus Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human Papillomavirus Vaccine (Experimental): The Gardasil HPV vaccine was administered in 3 doses: baseline, 2 months, and 6 months.
  Interventions: Biological: Human Papillomavirus Vaccine

INTERVENTIONS:
Biological: Human Papillomavirus Vaccine — 0.5mL intramuscular for 3 doses at 0, 2, and 6 months
  Other Names: Gardasil

SUMMARY:
The Gardasil vaccine, a vaccine targeted towards the human papillomavirus (HPV), has been shown to prevent the transmission of several strains of HPV in young women. Women with inflammatory bowel disease (IBD) may not respond as well to this vaccine, either due to having IBD or due to immunosuppressants used to control IBD. This study will test how well women with IBD respond to the Gardasil vaccine.

DETAILED DESCRIPTION:
Although guidelines exist for immunization of patients with inflammatory bowel disease, few studies exist demonstrating vaccine efficacy in this population. In patients with inflammatory bowel disease, lower than normal humoral responses have been shown with the tetanus toxoid booster, oral cholera, and influenza vaccinations. It is currently uncertain whether women with inflammatory bowel disease (IBD) have an increased risk of cervical dysplasia and cancer. Gardasil, a vaccine against human papilloma viruses (HPV) 6, 11, 16, and 18, has been approved for the prevention of cervical dysplasias and cancers in women ages 9-26 years. However, its immune response in immunocompromised or immunosuppressed patients is unknown.

Young women with inflammatory bowel disease who have not received the HPV vaccine will receive the vaccine. The vaccine is given in 3 doses over 6 months. Response to the vaccine will be measured 6 months after completing the vaccine series.

ELIGIBILITY:
Inclusion Criteria:

1. Women 9-26 years of age
2. Have inflammatory bowel disease (ie. Crohns disease or ulcerative colitis)

Exclusion Criteria:

1. Pregnancy
2. Taking corticosteroids
3. Allergy to yeast aluminum component of the HPV vaccine
4. Positive for all HPV types in the Gardasil vaccine-6, 11, 16, 18

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Tung, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2010 and January 2011, female patients between age 12-25 years of age were recruited through the Inflammatory Bowel Disease Clinics at the Mayo Clinic.
Period: Overall Study
Arm/Group | Human Papillomavirus Vaccine
Started | 15
Completed | 13 (One patient was found after enrollment to have already received one prior dose of the HPV vaccine.)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Human Papillomavirus Vaccine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 8
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 19.3 (3.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Disease Activity at First HPV vaccine dose [Number; unit: participants] — Participants were categorized as either having quiescent (inactivity or dormancy) or active disease activity at baseline, prior to first HPV vaccine dose.
  participants
    Quiescent | 9
    Active | 6

OUTCOME MEASURES:

1. Primary Outcome: Twelve Month Antibody Response to the Human Papillomavirus (HPV) Vaccine (Geometric Mean Titers [GMT])
Description: Anti-HPV levels were determined by an assay conducted by Merck & Co, Inc. and expressed as milliMerck units per milliliter (mMU/mL).
Time Frame: One year
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Human Papillomavirus Vaccine
Number analyzed (Participants) | 13
mMU/mL
  HPV 6 | 120.5 [69.3 to 209.4]
  HPV 11 | 175.0 [86.3 to 354.0]
  HPV 16 | 861.0 [559.8 to 1321.3]
  HPV 18 | 68.9 [34.9 to 135.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 12 month period of the study.
Arm/Group | Human Papillomavirus Vaccine
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 13/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Papillomavirus Vaccine (N=15)
Site reaction (Skin and subcutaneous tissue disorders) | 11 (11)
Malaise (General disorders) | 5 (5)
Headache (General disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Lightheadedness (General disorders) | 1 (1)
Sore Throat (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No